CLINICAL TRIAL: NCT06435390
Title: The Impact of the COVID-19 Pandemic on the Oral Hygiene Status of Children With High Caries Risk and Their Parents
Brief Title: Coronavirus Disease 2019 (COVID-19) Pandemic on the Oral Hygiene Status of Children
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Hanife ALTINIŞIK, Doç. Dr., Gazi University
Other Study IDs: E.630276
Record Dates: First submitted 2024-05-28; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: COVID-19 Pandemic
Keywords: COVID-19; oral hygiene; dietary habits; parents; pediatric dentistry
MeSH Terms: conditions — COVID-19; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3-5 year old 155 children with high caries risk and their parents: 3-5 year old 155 children with high caries risk and their parents before and after COVID-19

SUMMARY:
The purpose of this study is to compare oral hygiene status and dietary habits of 3-5 years old children and their parents with a questionnaire and clinic examination between pre- and post-COVID-19 period.

DETAILED DESCRIPTION:
Study Rationale and Objectives:

The primary motivation behind this study lies in understanding the impact of the COVID-19 pandemic on oral health behaviors, specifically focusing on children at high risk for dental caries.

Objectives include assessing changes in tooth brushing habits and dietary patterns among both children and their parents.

Study Design:

The study employs a prospective observational design. Participants are parents of 155 children aged 3-5 years. Data collection occurs at two time points: before and after the COVID-19 pandemic.

Data Collection Instruments:

A structured questionnaire is administered to parents. It covers:

Children's and parents' dietary habits (frequency of sugary food consumption). Oral hygiene practices (tooth brushing frequency). The index of decayed-missing-filled deciduous teeth (dmft) is used to assess dental caries status in children.

The COVID-19 pandemic had a limited impact on high-caries-risk children's tooth brushing habits.

However, increased sugary food consumption by both children and parents exacerbated caries risk.

Collaborative efforts between healthcare professionals and parents are crucial to mitigate negative oral health effects during such challenging times.

ELIGIBILITY:
Inclusion Criteria:

* 3-5 year old children with high caries risk. To identify high caries-risk children, the criteria used by the the American Academy of Pediatric Dentistry (AAPD) for assessing a child's dental caries risk were applied.

Exclusion Criteria:

* Childrens with systemic health problems and childrens with any space maintainers.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study used retrospective information for healthy 3-5 year old children with high caries risk and their parents who applied to the our University Pediatric Dentistry clinic between September 2019 and March 2020 (in the last six months before COVID-19)
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Changing tooth brushing and diet habits during the COVID-19 pandemic | from 15 March to 15 May 2022
  Changing tooth brushing and diet habits of 155 children aged 3-5 with high risk of caries during the COVID-19 pandemic period

CONTACTS AND LOCATIONS:
Overall Officials: ZELIHA HATİPOĞLU PALAZ, Principal Investigator — Gazi University; NAGEHAN AKTAŞ, Principal Investigator — Gazi University
Locations (1):
- Zeliha Hatipoğlu Palaz, Ankara, Biskek Street/ Emek, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Docimo R, Costacurta M, Gualtieri P, Pujia A, Leggeri C, Attina A, Cinelli G, Giannattasio S, Rampello T, Di Renzo L. Cariogenic Risk and COVID-19 Lockdown in a Paediatric Population. Int J Environ Res Public Health. 2021 Jul 15;18(14):7558. doi: 10.3390/ijerph18147558. PMID 34300008
- [Background] Gotler M, Oren L, Spierer S, Yarom N, Ashkenazi M. The impact of COVID-19 lockdown on maintenance of children's dental health: A questionnaire-based survey. J Am Dent Assoc. 2022 May;153(5):440-449. doi: 10.1016/j.adaj.2021.10.004. Epub 2021 Oct 19. PMID 35221097
- [Background] Mohapatra RK, Pintilie L, Kandi V, Sarangi AK, Das D, Sahu R, Perekhoda L. The recent challenges of highly contagious COVID-19, causing respiratory infections: Symptoms, diagnosis, transmission, possible vaccines, animal models, and immunotherapy. Chem Biol Drug Des. 2020 Nov;96(5):1187-1208. doi: 10.1111/cbdd.13761. Epub 2020 Jul 26. PMID 32654267
- [Background] Daly J, Black EAM. The impact of COVID-19 on population oral health. Community Dent Health. 2020 Nov 30;37(4):236-238. doi: 10.1922/CDH_Dec20editorialDalyBlack03. PMID 33269826
- [Background] Greuter W. [Practical industrial medicine in Switzerland]. Soz Praventivmed. 1981 Jul;26(3):126-9. doi: 10.1007/BF02081368. German. PMID 7293495
- [Background] Bonneau JC. [Contact allergy to sulfites: contact allergens, sources of exposure, and clinical profile]. Allerg Immunol (Paris). 1994 Nov;26(9):324-6. French. PMID 7865116
- [Background] Blumer S, Dagon N, Peretz B, Ratson T, Kharouba J. Function of the Family Unit, Oral Hygiene Rules and Attitudes to Dental Health in Children During First-Wave 2020 COVID-19 Lockdown. J Clin Pediatr Dent. 2021 Jan 1;45(1):1-7. doi: 10.17796/1053-4625-45.1.1. PMID 33690823
- [Background] Angelopoulou MV, Seremidi K, Papaioannou W, Gizani S. Impact of the COVID-19 lockdown on the oral health status of paediatric dental patients in Greece. Int J Paediatr Dent. 2023 May;33(3):246-253. doi: 10.1111/ipd.13048. Epub 2023 Mar 13. PMID 36680387
- [Background] Goswami M, Grewal M, Garg A. Attitude and practices of parents toward their children's oral health care during COVID-19 pandemic. J Indian Soc Pedod Prev Dent. 2021 Jan-Mar;39(1):22-28. doi: 10.4103/jisppd.jisppd_478_20. PMID 33885383
- [Background] Mahagna M, Nir I, Larbier M, Nitsan Z. Effect of age and exogenous amylase and protease on development of the digestive tract, pancreatic enzyme activities and digestibility of nutrients in young meat-type chicks. Reprod Nutr Dev. 1995;35(2):201-12. doi: 10.1051/rnd:19950208. PMID 7537505
- [Background] Dickson-Swift V, Kangutkar T, Knevel R, Down S. The impact of COVID-19 on individual oral health: a scoping review. BMC Oral Health. 2022 Sep 22;22(1):422. doi: 10.1186/s12903-022-02463-0. PMID 36138456
- [Background] Navarro-Perez CF, Fernandez-Aparicio A, Gonzalez-Jimenez E, Montero-Alonso MA, Schmidt-RioValle J. Effects of COVID-19 lockdown on the dietary habits and lifestyle in a population in southern Spain: a cross-sectional questionnaire. Eur J Clin Nutr. 2022 Jun;76(6):883-890. doi: 10.1038/s41430-021-01034-w. Epub 2021 Oct 28. PMID 34711931
- [Background] Olszewska A, Paszynska E, Roszak M, Czajka-Jakubowska A. Management of the Oral Health of Children During the COVID-19 Pandemic in Poland. Front Public Health. 2021 Jul 29;9:635081. doi: 10.3389/fpubh.2021.635081. eCollection 2021. PMID 34395353
- [Background] Tellez M, Gomez J, Pretty I, Ellwood R, Ismail AI. Evidence on existing caries risk assessment systems: are they predictive of future caries? Community Dent Oral Epidemiol. 2013 Feb;41(1):67-78. doi: 10.1111/cdoe.12003. PMID 22978796
- [Background] Costa AL, Pereira JL, Franco L, Guinot F. COVID-19 Lockdown: Impact on Oral Health-Related Behaviors and Practices of Portuguese and Spanish Children. Int J Environ Res Public Health. 2022 Nov 30;19(23):16004. doi: 10.3390/ijerph192316004. PMID 36498079
- [Background] Caramida M, Dumitrache MA, Tancu AMC, Ilici RR, Ilinca R, Sfeatcu R. Oral Habits during the Lockdown from the SARS-CoV-2 Pandemic in the Romanian Population. Medicina (Kaunas). 2022 Mar 5;58(3):387. doi: 10.3390/medicina58030387. PMID 35334563
- [Background] Ruiz-Roso MB, de Carvalho Padilha P, Mantilla-Escalante DC, Ulloa N, Brun P, Acevedo-Correa D, Arantes Ferreira Peres W, Martorell M, Aires MT, de Oliveira Cardoso L, Carrasco-Marin F, Paternina-Sierra K, Rodriguez-Meza JE, Montero PM, Bernabe G, Pauletto A, Taci X, Visioli F, Davalos A. Covid-19 Confinement and Changes of Adolescent's Dietary Trends in Italy, Spain, Chile, Colombia and Brazil. Nutrients. 2020 Jun 17;12(6):1807. doi: 10.3390/nu12061807. PMID 32560550
- [Background] Hamilton K, Cornish S, Kirkpatrick A, Kroon J, Schwarzer R. Parental supervision for their children's toothbrushing: Mediating effects of planning, self-efficacy, and action control. Br J Health Psychol. 2018 May;23(2):387-406. doi: 10.1111/bjhp.12294. Epub 2018 Jan 18. PMID 29349924
- [Background] Kotha SB, AlFaraj NSM, Ramdan TH, Alsalam MA, Al Ameer MJ, Almuzin ZM. Associations between Diet, Dietary and Oral Hygiene Habits with Caries Occurrence and Severity in Children with Autism at Dammam City, Saudi Arabia. Open Access Maced J Med Sci. 2018 Jun 6;6(6):1104-1110. doi: 10.3889/oamjms.2018.245. eCollection 2018 Jun 20. PMID 29983812
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/34300008/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/35221097/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/32654267/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/33269826/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/32569870/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/33549091/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/33690823/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/36680387/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/33885383/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/32978848/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/36138456/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/34711931/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/34395353/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/22978796/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/36498079/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/35334563/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/32560550/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/29349924/
- See also: COVID-19 Pandemic — http://pubmed.ncbi.nlm.nih.gov/29983812/